CLINICAL TRIAL: NCT05192564
Title: Supervised Exercise as an Adjuvant Program in People With Chronic Bilateral or Unilateral Vestibular Hypofunction: EXERVEST Study
Brief Title: Exercise and Vestibular Hypofunction
Acronym: EXERVEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: Bioaraba (Unknown)
Responsible Party: Principal Investigator, SARA MALDONADO-MARTIN, Principal Investigator, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXERcise+VESTibular (EXERVEST)
Record Dates: First submitted 2021-11-25; First posted 2022-01-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Vestibular Disease; Vestibular Disorder; Vestibular Vertigo
Keywords: Vestibular hypofunction; Exercise; Balance training; Imbalance
MeSH Terms: conditions — Vestibular Diseases; Vertigo; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: DESIGN: Controlled, randomized, prospective, single-blind (staff of the otorhinolaryngology department) intervention study carried out in a cohort of patients (over 18 yr old) with a diagnosis of bilateral or unilateral vestibular hypofunction divided into two groups: intervention group with exercise + conventional rehabilitation treatment (EX group) and a group without intervention that will receive only conventional rehabilitation treatment (attention control group, AC).
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EX Group (Experimental): Conventional rehabilitation treatment plus exercise intervention under the supervision of exercise specialists two non-consecutive days per week for eight weeks.
  Interventions: Other: Exercise for bilateral or unilateral vestibular hypofunction patients; Other: Conventional rehabilitation treatment
- AC Group - ATTENTION CONTROL GROUP (Active Comparator): Conventional rehabilitation treatment at home with unsupervised exercise intervention
  Interventions: Other: Conventional rehabilitation treatment

INTERVENTIONS:
Other: Exercise for bilateral or unilateral vestibular hypofunction patients — Physical Activity intervention with balance exercises, multidirectional displacements, and strength with postural control, implementing 8-10 exercises integrating the main muscle groups and motor patterns, aerobic exercise on bicycle (15 min) developed progressively in intensity (R1-mild, R2-moderate, R3-vigorous) implementing an intervallic design in low volume.
  Arms: EX Group
Other: Conventional rehabilitation treatment — Vestibular rehabilitation exercises counseling

SUMMARY:
Vestibular hypofunction is a heterogeneous clinical entity that arises after a vestibular pathway injury, which if not properly compensated becomes chronic, and very often disabling, presenting with postural instability, blurred vision with cephalic movement, oscillopsia, and subjective sensation of dizziness and imbalance. People diagnosed with vestibular hypofunction, because of their clinical condition, often tend to reduce physical activity and lead to a sedentary life, despite the fact that exercise has been shown to improve postural stability, and it is a determining factor in recovery after vestibular injury. Physical activity improves the quality of life and reduces the risk of falls. Supervised exercise is, therefore, among the potentially beneficial adjuvant programs in this population, although little has been studied in comparison with other pathologies. Furthermore, in vestibular hypofunction, there is insufficient evidence on specific interventions in specific clinical situations, the amount of exercise, and the optimal duration of the programs. Therefore, the aims of the study are 1) to analyze the effects on balance by an 8-week period of a supervised exercise program in people with a diagnosis of bilateral or unilateral vestibular hypofunction and 2) to examine the effect of six-months detraining subsequent to intervention. Secondary objectives are to examine the additional effect of the intervention on health-related quality of life, psychological well-being, cardiorespiratory fitness, body composition, blood pressure, physical activity level, sedentary behavior, and sleep quality.

DETAILED DESCRIPTION:
Interventional study with two randomized groups (attention control '[AC] and exercise group,[EX]) with assessment pre and post-intervention (8 weeks) and 6 months follow-up.

The AC group will perform only the home vestibular rehabilitation exercises that are usually prescribed in consultation with this type of patient, performing the same assessments as the intervention group in all phases of the study.

The participants in the EX group will exercise under the supervision of specialists in exercise and sports physical educators two non-consecutive days per week for eight weeks at the Faculty of Education and Sport of the University of the Basque Country (UPV/EHU). All sessions will start and end with blood pressure measurements and exercise intensity will be monitored by heart rate monitors (Polar Electro, Kempele, Finland) and through the original Borg scale (6-20). All sessions will include a 5-10 min warm-up with joint mobility exercises and gait technique and a 10 min cooldown with basic stretching exercises and controlled breathing. The main part of the session will consist of: 1) balance exercises, multidirectional displacements and strength with postural control, implementing 8-10 exercises integrating the main muscle groups and motor patterns, 2) aerobic exercise on bicycle (15 min) developed progressively in intensity (R1-mild, R2-moderate, R3-vigorous) implementing an intervallic design at low volume. The physical exercise intensity ranges (R1-mild, R2-moderate, R3-vigorous) will be defined on an individualized basis from the initial stress test and based on ventilatory thresholds. At the end of the intervention, participants will be provided with information on physical activity recommendations. Both intervention and control group patients will have all antivertiginous drugs withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Patient with bilateral or unilateral vestibular hypofunction.
* More than 6 months since the onset of vestibular hypofunction (chronic instability).
* Age over 18 years old.
* No previous rehabilitation treatment for vestibular hypofunction other than home exercises.

Exclusion Criteria:

* Fluctuating instability (not present every day).
* Recent onset instability (less than 6 months old, susceptible to complete clinical recovery).
* Current neurological pathology.
* History of neurosurgical disease, cerebrovascular disease, neurodegenerative disease or with central nervous system sequelae.
* Uncorrected ocular disorders.
* History of peripheral neuropathy in the lower extremities.
* Arthropathy or motor defects in lower limbs.
* Prolonged use of sedatives or vestibular suppressant medication.
* Significant medical disorders: including uncontrolled arterial hypertension, chronic or recurrent respiratory, neuromuscular or psychiatric diseases; musculoskeletal problems that interfere with physical exercise; immunodeficient diseases or a positive HIV test; anemia, blood disorders, chronic thrombotic disorders or hypercoagulant states; malignant tumors within the last five years, with the exception of therapeutically controlled skin cancer; any other disease that may be affected or aggravated by physical exercise.
* Being pregnant or breastfeeding.
* Have plans to be out of town for more than two weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-01-08 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Balance | 8-week time
  Computerized Dynamic Posturography testing can objectively measure a patient's three sensory inputs at one time during the Sensory Oorganization Test. It can provide insight into where the balance disturbance may be developing from and more importantly, which one of the sensory inputs shows a problem. The human body uses three sensory inputs to maintain balance proper balance, they are: Vestibular (inner ear system), Somatosenory (feet, ankles, joints), Vision (eyes). These sensory inputs interact with the brain, which then drive and control our motor functions. Computerized Dynamic Posturography is a unique assessment technique used to objectively quantify and differentiate among these three sensory inputs, along with motor, and central adaptive impairments to balance control.

SECONDARY OUTCOMES:
Health-related Quality of life | 8-week time
  Measured by Dizziness Handicap Inventory Questionnaire It contains a total score (100 items) and scores in the physical (28 items), functional (36 items) and emotional (36 items) subscales.
  Scores greater than 10 points should be referred to balance specialists for further evaluation.
  16-34 Points (mild handicap) 36-52 Points (moderate handicap) 54+ Points (severe handicap)
Depression | 8-week time
  Measured by Beck Depression Inventory (BDI) 21 Likert-type items. The maximum score is 63 points, with the following classification: 0-13, minimal depression; 14-19, mild depression; 20-28, moderate depression; and 29-63, severe depression.
Physical activity level | 8-week time
  Measured by accelerometry (8 days) in the non-dominant wrist.
Blood pressure | 8-week time
  Ambulatory blood pressure monitoring (AMBP) is accomplished with a special device that consists of a blood pressure cuff that is worn on the arm and is attached to a small recording device that you wear on your belt. The participant will wear the ABPM device for 24 hours, and it records your blood pressure periodically (30-min intervals) throughout that period, during your routine daily activities and while you are sleeping.
Body composition | 8-week time
  Biolectrical impedance for estimating % of body fat-mass, muscle-mass, and water.
Cardiorespiratory fitness | 8-week time
  Peak Cardiopulmonary exercise test on bicycle ergometer.
Anxiety | 8-week time
  Beck Anxiety Inventory (BAI). 21 items. The maximum score is 63 points, 25.7±11.4 being considered an anxiety score.
Physical activity and sedentary behaviour | 8-week time
  International physical activity questionnaire (IPAQ) short-version. It consists of seven questions to capture average daily time spent sitting, walking, and engaging in moderate and vigorous PA over the last seven days.
Assessment of gait, balance and risk of falls | 8-week time
  Dynamic Gait Index (DGI): composed of 8 exercises each scored from 0 (severe impairment) to 3 (highest level of functionality); maximum score: 24 points; a score < 19 is predictive of falls.
Waist circumference | 8-week time
  Stand and place a tape measure around your middle, just above your hipbones. Measured in cm
Body mass index (BMI) | 8-week time
  BMI is a person's weight in kilograms divided by the square of height in meters.

CONTACTS AND LOCATIONS:
Overall Officials: SARA MALDONADO-MARTIN, PhD, Principal Investigator — University of the Basque Country (UPV/EHU)
Locations (1):
- Faculty of Education and Sport, Vitoria-Gasteiz, Basque Country, Spain

REFERENCES:
- [Background] Strupp M, Kim JS, Murofushi T, Straumann D, Jen JC, Rosengren SM, Della Santina CC, Kingma H. Bilateral vestibulopathy: Diagnostic criteria Consensus document of the Classification Committee of the Barany Society. J Vestib Res. 2017;27(4):177-189. doi: 10.3233/VES-170619. PMID 29081426
- [Background] Grill E, Heuberger M, Strobl R, Saglam M, Holle R, Linkohr B, Ladwig KH, Peters A, Schneider E, Jahn K, Lehnen N. Prevalence, Determinants, and Consequences of Vestibular Hypofunction. Results From the KORA-FF4 Survey. Front Neurol. 2018 Dec 7;9:1076. doi: 10.3389/fneur.2018.01076. eCollection 2018. PMID 30581415
- [Background] Morimoto H, Asai Y, Johnson EG, Koide Y, Niki J, Sakai S, Nakayama M, Kabaya K, Fukui A, Mizutani Y, Mizutani T, Ueki Y, Mizutani J, Ueki T, Wada I. Objective measures of physical activity in patients with chronic unilateral vestibular hypofunction, and its relationship to handicap, anxiety and postural stability. Auris Nasus Larynx. 2019 Feb;46(1):70-77. doi: 10.1016/j.anl.2018.06.010. Epub 2018 Jun 30. PMID 30691599
- [Background] Starkov D, Strupp M, Pleshkov M, Kingma H, van de Berg R. Diagnosing vestibular hypofunction: an update. J Neurol. 2021 Jan;268(1):377-385. doi: 10.1007/s00415-020-10139-4. Epub 2020 Aug 7. PMID 32767115
- [Background] van Esch BF, Nobel-Hoff GE, van Benthem PP, van der Zaag-Loonen HJ, Bruintjes TD. Determining vestibular hypofunction: start with the video-head impulse test. Eur Arch Otorhinolaryngol. 2016 Nov;273(11):3733-3739. doi: 10.1007/s00405-016-4055-9. Epub 2016 Apr 25. PMID 27113255
- [Background] Visser JE, Carpenter MG, van der Kooij H, Bloem BR. The clinical utility of posturography. Clin Neurophysiol. 2008 Nov;119(11):2424-36. doi: 10.1016/j.clinph.2008.07.220. Epub 2008 Sep 12. PMID 18789756
- [Background] Hillier S, McDonnell M. Is vestibular rehabilitation effective in improving dizziness and function after unilateral peripheral vestibular hypofunction? An abridged version of a Cochrane Review. Eur J Phys Rehabil Med. 2016 Aug;52(4):541-56. Epub 2016 Jul 12. PMID 27406654
- [Background] Sulway S, Whitney SL. Advances in Vestibular Rehabilitation. Adv Otorhinolaryngol. 2019;82:164-169. doi: 10.1159/000490285. Epub 2019 Jan 15. PMID 30947180
- [Background] Kundakci B, Sultana A, Taylor AJ, Alshehri MA. The effectiveness of exercise-based vestibular rehabilitation in adult patients with chronic dizziness: A systematic review. F1000Res. 2018 Mar 5;7:276. doi: 10.12688/f1000research.14089.1. eCollection 2018. PMID 29862019
- [Background] Hall CD, Herdman SJ, Whitney SL, Cass SP, Clendaniel RA, Fife TD, Furman JM, Getchius TS, Goebel JA, Shepard NT, Woodhouse SN. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Evidence-Based Clinical Practice Guideline: FROM THE AMERICAN PHYSICAL THERAPY ASSOCIATION NEUROLOGY SECTION. J Neurol Phys Ther. 2016 Apr;40(2):124-55. doi: 10.1097/NPT.0000000000000120. PMID 26913496
- [Background] Dunlap PM, Holmberg JM, Whitney SL. Vestibular rehabilitation: advances in peripheral and central vestibular disorders. Curr Opin Neurol. 2019 Feb;32(1):137-144. doi: 10.1097/WCO.0000000000000632. PMID 30461465
- [Background] Maslovara S, Butkovic-Soldo S, Peric M, Pajic Matic I, Sestak A. Effect of vestibular rehabilitation on recovery rate and functioning improvement in patients with chronic unilateral vestibular hypofunction and bilateral vestibular hypofunction. NeuroRehabilitation. 2019;44(1):95-102. doi: 10.3233/NRE-182524. PMID 30776020
- [Background] Meldrum D, Jahn K. Gaze stabilisation exercises in vestibular rehabilitation: review of the evidence and recent clinical advances. J Neurol. 2019 Sep;266(Suppl 1):11-18. doi: 10.1007/s00415-019-09459-x. Epub 2019 Aug 5. PMID 31385017
- [Background] Viziano A, Micarelli A, Augimeri I, Micarelli D, Alessandrini M. Long-term effects of vestibular rehabilitation and head-mounted gaming task procedure in unilateral vestibular hypofunction: a 12-month follow-up of a randomized controlled trial. Clin Rehabil. 2019 Jan;33(1):24-33. doi: 10.1177/0269215518788598. Epub 2018 Jul 16. PMID 30012022
- [Background] Arnold SA, Stewart AM, Moor HM, Karl RC, Reneker JC. The Effectiveness of Vestibular Rehabilitation Interventions in Treating Unilateral Peripheral Vestibular Disorders: A Systematic Review. Physiother Res Int. 2017 Jul;22(3). doi: 10.1002/pri.1635. Epub 2015 Jun 25. PMID 26111348
- [Background] Balaban CD, Hoffer ME, Gottshall KR. Top-down approach to vestibular compensation: translational lessons from vestibular rehabilitation. Brain Res. 2012 Oct 30;1482:101-11. doi: 10.1016/j.brainres.2012.08.040. Epub 2012 Sep 6. PMID 22981400
- [Background] Yardley L, Redfern MS. Psychological factors influencing recovery from balance disorders. J Anxiety Disord. 2001 Jan-Apr;15(1-2):107-19. doi: 10.1016/s0887-6185(00)00045-1. PMID 11388354
- [Background] Ekwall A, Lindberg A, Magnusson M. Dizzy - why not take a walk? Low level physical activity improves quality of life among elderly with dizziness. Gerontology. 2009;55(6):652-9. doi: 10.1159/000235812. Epub 2009 Aug 25. PMID 19707007
- [Background] Smolka W, Smolka K, Markowski J, Pilch J, Piotrowska-Seweryn A, Zwierzchowska A. The efficacy of vestibular rehabilitation in patients with chronic unilateral vestibular dysfunction. Int J Occup Med Environ Health. 2020 Apr 30;33(3):273-282. doi: 10.13075/ijomeh.1896.01330. Epub 2020 Mar 26. PMID 32235946
- [Background] Jahn K, Lopez C, Zwergal A, Zur O, Cakrt O, Kellerer S, Kerkeni H, Tjernstrom F, Meldrum D; Vestibular Rehabilitation Research Group in the European DIZZYNET. Vestibular rehabilitation therapy in Europe: chances and challenges. J Neurol. 2019 Sep;266(Suppl 1):9-10. doi: 10.1007/s00415-019-09368-z. Epub 2019 May 17. No abstract available. PMID 31102020
- [Derived] Ruiz-Rios M, Lekue A, Pinedo-Lopez J, Tous-Espelosin M, Arratibel-Imaz I, Garcia-Tabar I, Maldonado-Martin S. Supervised multicomponent exercise as an adjuvant program for people with unilateral and/or bilateral chronic vestibular hypofunction: EXERVEST study protocol. Contemp Clin Trials Commun. 2023 Oct 6;36:101213. doi: 10.1016/j.conctc.2023.101213. eCollection 2023 Dec. PMID 37868660